CLINICAL TRIAL: NCT04941560
Title: Artificial Intelligence to Assess the Association Between Multi-dimension Facial Characteristics and Coronary Artery Diseases
Brief Title: Assessing the Association Between Multi-dimension Facial Characteristics and Coronary Artery Diseases
Status: Completed | Type: Observational
Sponsor: China National Center for Cardiovascular Diseases (Other Government)
Responsible Party: Sponsor
Other Study IDs: 20210621-2021-1471
Record Dates: First submitted 2021-06-22; First posted 2021-06-28 (Actual); Last update posted 2023-03-21 (Actual); Status verified 2023-03

CONDITIONS: Coronary Artery Disease
Keywords: Artificial intelligence; Facial characteristics
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Algorithm training and test group: Patients undergoing coronary angiography or coronary computer tomography angiography will be enrolled. Patients data will be used to training and validate the algorithm for CAD detection based on facial photos.
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — No intervention

SUMMARY:
The purposes of this study are 1) to explore the association between multi-dimension facial characteristics and the increased risk of coronary artery diseases (CAD); 2) to evaluate the diagnostic efficacy of multi-dimension appearance factors for coronary artery diseases.

DETAILED DESCRIPTION:
Previous study demonstrated the feasibility of using deep learning to detect coronary artery disease based on facial photos. However, several limitations made the algorithm hard to be utilized in clinical practice, including low specificity and lack of external validation. Adding multi-dimension facial characteristics may further increase the algorithm effect.

Thus, the investigators designed a single-center, cross-sectional study to explore the association between multi-dimension facial characteristics and CAD and to evaluate the predictive efficacy of multi-dimension appearance factors for CAD. The investigators will recruit patients undergoing coronary angiography or coronary computer tomography angiography. Patients' baseline information and multi-dimension facial images will be collected. The investigators will train and validate a deep learning algorithm based on multi-dimension facial photos.

ELIGIBILITY:
Inclusion Criteria:

* Undergoing coronary angiography or coronary computer tomography angiography
* Written informed consent

Exclusion Criteria:

* Prior percutaneous coronary intervention (PCI)
* Prior coronary artery bypass graft (CABG)
* Screening coronary artery disease before treating other heart diseases
* Without blood biochemistry outcome
* With artificially facial alteration (i.e. cosmetic surgery, facial trauma or make-up)
* Other situations which make patients fail to be photographed

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients who undergo coronary angiography or coronary computer tomography angiography from both resident patients and outpatient.
Sampling Method: Non-Probability Sample
Enrollment: 460 (Actual)
Dates: Start 2021-09-06 (Actual); Primary Completion 2023-02-10 (Actual); Study Completion 2023-02-10 (Actual)

PRIMARY OUTCOMES:
Area under receiver operating curve (AUC) | At the end of enrollment (1 mouth)
  Area under receiver operating curve of algorithm assessed in test group

SECONDARY OUTCOMES:
Sensitivity of algorithm | At the end of enrollment (1 mouth)
  Sensitivity of algorithm assessed in test group
Specificity of algorithm | At the end of enrollment (1 mouth)
  Specificity of algorithm assessed in test group
Positive predictive value (PPV) | At the end of enrollment (1 mouth)
  PPV of algorithm assessed in test group
Negative predictive value (NPV) | At the end of enrollment (1 mouth)
  NPV of algorithm assessed in test group
Diagnostic accuracy rate | At the end of enrollment (1 mouth)
  Diagnostic accuracy rate of algorithm assessed in test group

CONTACTS AND LOCATIONS:
Locations (1):
- Fuwai hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No